CLINICAL TRIAL: NCT06312267
Title: Reducing Wound Infections Using Bioelectric Wound Dressings
Acronym: JumpStart
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1840655
Record Dates: First submitted 2024-03-07; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Surgical Site Infection
Keywords: Surgery outcomes; Bioelectric dressing,
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: Total of 20 patients will be identified and divided in two groups (control and experimental group). 10 of the patients undergo surgery using current ERAS protocol standard of care skin cleaning preparation. The other 10 patients skin prep will be substituted with the Bioelectrical dressing preoperatively and post-operative.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control Arm (No Intervention): Study participants will undergo surgery using current ERAS protocol standard of care skin cleaning preparation.
- Experimental Arm (Experimental): Study participants will use Bioelectrical dressing preoperatively and post-operative.
  Interventions: Device: Bioelectric dressing

INTERVENTIONS:
Device: Bioelectric dressing — Participants randomized into the experimental arm will have a bioelectric dressing applied 3 days before surgery, and 3 days post-surgery.
  Arms: Experimental Arm

SUMMARY:
The purpose of this study is to compare the outcomes of using Bioelectric wound dressing on the pre-operative wound site and post operatively and compared it outcomes to the standard of care chlorhexidine skin preparation.

DETAILED DESCRIPTION:
The standard of care for enhance recovery after surgery (ERAS) protocol uses chlorhexidine alcohol base prep as the way to clean the skin preoperatively to decrease bacterial flora before sterile prep at the OR.

Under ERAS protocol there is no recommendations on any post-operative dressing. Biolelectric wound dressing has been introduced, used and proof to decrease wound infection in orthopedic extremity clean surgery for years.

The purpose of this study is to compare the outcomes of using Bioelectric wound dressing on the pre-operative wound site and post operatively and compared it outcomes to the standard of care chlorhexidine skin preparation.

ELIGIBILITY:
Inclusion Criteria:

1. Elective diverticular, benign polyp, or colon cancer resection
2. Age 18-90 years old
3. All patients must receive some kind of bowel prep (SU- prep, pills, Go-Lytely, milk of magnesia, etc.…)
4. Must be off antibiotics for more than 2 weeks before surgery
5. Surgery must be laparoscopic, hand assisted or Robotic
6. Skin will be closed in layers and subcuticular interrupted fashion
7. Just one dose of preoperative antibiotics (Invanz or equivalent if patient is allergic)
8. Patients will have a primary anastomosis, no colostomy.
9. Patient must be compliant with dressing care
10. Ability to provide informed consent

Exclusion Criteria:

1. Active infections before surgery -example: Intra-abdominal abscess not drained or actively on antibiotics on the day of surgery, skin infections
2. Inability to take intestinal bowel preparation
3. HgbA1c >8
4. BMI >40
5. Immunosuppression
6. Need of steroid stress dose pre-op
7. Patient receiving active chemotherapy
8. Need of stoma (end ostomies after resection protective stoma included)
9. Need of blood transfusion during surgery
10. Use of irrigation with antibiotics or IRRISEPTR during surgery
11. Any standard contraindication to anesthesia and/or surgery
12. Pregnancy or lactating women
13. Inability to provide informed consent
14. Inability to follow instructions for dressing care
15. Sensitivity or allergy to silver or zinc

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Quantitative bacterial count | 4 total biopsies will be collected. (3 days before surgery, surgery day pre incision, immediately post-surgery and 3 days post-surgery)
  Skin biopsies will be collected and analyzed for bacterial counts

CONTACTS AND LOCATIONS:
Overall Officials: Jay Redan, MD, Principal Investigator — AdventHealth
Locations (1):
- AdventHealth Celebration, Kissimmee, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gustafsson UO, Scott MJ, Hubner M, Nygren J, Demartines N, Francis N, Rockall TA, Young-Fadok TM, Hill AG, Soop M, de Boer HD, Urman RD, Chang GJ, Fichera A, Kessler H, Grass F, Whang EE, Fawcett WJ, Carli F, Lobo DN, Rollins KE, Balfour A, Baldini G, Riedel B, Ljungqvist O. Guidelines for Perioperative Care in Elective Colorectal Surgery: Enhanced Recovery After Surgery (ERAS(R)) Society Recommendations: 2018. World J Surg. 2019 Mar;43(3):659-695. doi: 10.1007/s00268-018-4844-y. PMID 30426190
- [Background] Cooke CL, Greene RS, van Eck CF, Uquilas C, Limpisvasti O. Bioelectric Silver-Zinc Dressing Equally Effective to Chlorhexidine in Reducing Skin Bacterial Load in Healthy Volunteers. Arthroscopy. 2018 Oct;34(10):2886-2891. doi: 10.1016/j.arthro.2018.05.046. Epub 2018 Sep 5. PMID 30195951
- [Background] Kim H, Park S, Housler G, Marcel V, Cross S, Izadjoo M. An Overview of the Efficacy of a Next Generation Electroceutical Wound Care Device. Mil Med. 2016 May;181(5 Suppl):184-90. doi: 10.7205/MILMED-D-15-00157. PMID 27168571
- [Background] Banerjee J, Das Ghatak P, Roy S, Khanna S, Hemann C, Deng B, Das A, Zweier JL, Wozniak D, Sen CK. Silver-zinc redox-coupled electroceutical wound dressing disrupts bacterial biofilm. PLoS One. 2015 Mar 24;10(3):e0119531. doi: 10.1371/journal.pone.0119531. eCollection 2015. PMID 25803639
- [Background] Banerjee J, Das Ghatak P, Roy S, Khanna S, Sequin EK, Bellman K, Dickinson BC, Suri P, Subramaniam VV, Chang CJ, Sen CK. Improvement of human keratinocyte migration by a redox active bioelectric dressing. PLoS One. 2014 Mar 3;9(3):e89239. doi: 10.1371/journal.pone.0089239. eCollection 2014. PMID 24595050
- [Background] Barki KG, Das A, Dixith S, Ghatak PD, Mathew-Steiner S, Schwab E, Khanna S, Wozniak DJ, Roy S, Sen CK. Electric Field Based Dressing Disrupts Mixed-Species Bacterial Biofilm Infection and Restores Functional Wound Healing. Ann Surg. 2019 Apr;269(4):756-766. doi: 10.1097/SLA.0000000000002504. PMID 29099398
- [Background] Kim H, Makin I, Skiba J, Ho A, Housler G, Stojadinovic A, Izadjoo M. Antibacterial efficacy testing of a bioelectric wound dressing against clinical wound pathogens. Open Microbiol J. 2014 Feb 21;8:15-21. doi: 10.2174/1874285801408010015. eCollection 2014. PMID 24627730
- [Background] Kim H, Izadjoo MJ. Antibiofilm efficacy evaluation of a bioelectric dressing in mono- and multi-species biofilms. J Wound Care. 2015 Feb;24 Suppl 2:S10-4. doi: 10.12968/jowc.2015.24.Sup2.S10. PMID 25647504
- [Background] Kulkarni N, Arulampalam T. Laparoscopic surgery reduces the incidence of surgical site infections compared to the open approach for colorectal procedures: a meta-analysis. Tech Coloproctol. 2020 Oct;24(10):1017-1024. doi: 10.1007/s10151-020-02293-8. Epub 2020 Jul 9. PMID 32648141
- [Result] Hubner M, Diana M, Zanetti G, Eisenring MC, Demartines N, Troillet N. Surgical site infections in colon surgery: the patient, the procedure, the hospital, and the surgeon. Arch Surg. 2011 Nov;146(11):1240-5. doi: 10.1001/archsurg.2011.176. Epub 2011 Jul 18. PMID 21768407